CLINICAL TRIAL: NCT01319747
Title: Video-Assisted Thoracoscopic Pulmonary Vein Isolation Versus Percutaneous Catheter Ablation in Atrial Fibrillation Trial
Acronym: VATCAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion rate insufficient
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, B. Oude Velthuis, B. Oude Velthuis MD, Medisch Spectrum Twente
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL32865.044.10; 32865 (Other: CCMO ABR Nummer); Dutch trial register entry (Registry Identifier: NTR2455)
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial; fibrillation; pvi; vats; ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous therapy (Active Comparator)
  Interventions: Procedure: PVI
- VATS therapy (Active Comparator)
  Interventions: Procedure: VATS-PVI

INTERVENTIONS:
Procedure: PVI — For catheter ablation, we used irrigated 4mm RF-ablation catheters, at a maximum power of 30-35Watt, an irrigation rate of 20 mL/min. PV isolation was performed by wide circumferential ablation, encircling all ipsilateral PVs.
  Arms: Percutaneous therapy
Procedure: VATS-PVI — A bilateral video-assisted thoracoscopic (VATS) pulmonary vein isolation and left atrial appendage (LAA) excision is performed under general anaesthesia and double-lumen endotracheal ventilation.
  Arms: VATS therapy

SUMMARY:
Recent studies demonstrated that radiofrequency isolation of the pulmonary veins (PVI) and surgically video assisted thorascopic pulmonary vein isolation (VATS-PVI) are acceptable or even superior alternatives to antiarrhythmic drug therapy in patients with symptomatically paroxysmal atrial fibrillation (AF). However, data comparing effectiveness in both interventions are limited.

The investigators want to compare the effectiveness of PVI and VATS-PVI. Secondary objectives are to compare the duration of hospitalization, quality of Life, cost and to compare the satisfaction of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Documented, symptomatic, episodes of paroxysmal or persistent AF
* During the last 6 months patients must have at least 2 documented episodes of AF, despite the use of at least 1 anti arrhythmic drug.
* Able of providing informed consent

Exclusion Criteria:

* Pregnancy
* Unwillingness to use or contra-indications for vitamin K antagonists
* Severely enlarged left atrium (>50 mm) on echocardiography
* Prior AF ablation or AF surgery
* Intracardiac thrombus
* Prior heart surgery or pulmonary disease hampering thoracoscopic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-09; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Recurrence of AF | one year
  The percentage of patients without a recurrence of AF, without antiarrhythmic drugs (AADs), within a follow-up period of at least 12 months after a stabilisation period of 90 days after the initial procedure. An episode of AF is defined as an episode of at least 30 seconds duration.

SECONDARY OUTCOMES:
Treatment impact | one year
  Secondary objectives include the duration and cost of hospitalization, discomfort during admission, assessment and experienced AF burden during follow-up of procedural impact on the patient and time to recurrence after intervention. A complication register will also be kept.

CONTACTS AND LOCATIONS:
Overall Officials: Marcoen Scholten, MD PhD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands